CLINICAL TRIAL: NCT04796324
Title: Phase II, Open Label, Single Arm Study to Investigate Anti-tumor Effect of Ixabepilone in Patients With Locally Recurrent or Metastatic Breast Cancer (mBC) Selected by the Ixabepilone DRP After Failure of an Anthracycline and Taxanes.
Brief Title: Anti-tumor Effect of Ixabepilone in Metastatic Breast Cancer (mBC) Selected by the Ixabepilone DRP.
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Allarity Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-2001
Record Dates: First submitted 2021-03-08; First posted 2021-03-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone

STUDY DESIGN:
Intervention Model Description: Ixabepilone 40 mg/m2 is administered as a 3-h intravenous infusion Day 1 in a 3-week cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixabepilone (Experimental): Ixabepilone 40 mg/m2 is administered as a 3-h intravenous infusion Day 1 in a 3-week cycle
  Interventions: Drug: Ixabepilone Injection

INTERVENTIONS:
Drug: Ixabepilone Injection — Ixabepilone 40 mg/m2 is administered as a 3-h intravenous infusion Day 1 in a 3-week cycle

SUMMARY:
The purpose is to investigate anti-tumor effect of ixabepilone in patients with locally recurrent or metastatic breast cancer (mBC) selected by the Ixabepilone DRP after failure of an anthracycline and taxanes.

DETAILED DESCRIPTION:
Patients will be screened with the Ixabepilone DRP. If the tumor tissue has a DRP( Drug Response Prediction) score of >67% (Belgium >33%) the patient can be included in the clinical study. Ixabepilone 40 mg/m2 is administered as a 3-h intravenous infusion Day 1 in a 3-week cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Age 18 years or older
3. Patients with histologically or cytological confirmed carcinoma of the breast. Patients with locally recurrent or metastatic disease
4. Patients with HR-positive, HER negative tumors or triple negative tumors
5. Previous chemotherapies (neo, adjuvant or in the metastatic setting) must have included a taxane and an anthracycline unless anthracycline therapy is not indicated.
6. Maximum of three (3) prior chemotherapies in the metastatic setting in addition to any number of prior lines of endocrine therapy
7. Measurable disease
8. Performance status of ECOG ≤ 1
9. With an Ixabepilone DRP - score of >33% (Germany >67%)
10. Adequate conditions as evidenced by the following clinical laboratory values:

    1. Absolute neutrophils count (ANC) ≥ 1.5 x 109/L
    2. Hemoglobin > 6.2 mmol/L
    3. Platelets ≥ 100 x 109 /L
    4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN
    5. Serum bilirubin ≤ 1.0 ULN
    6. Alkaline phosphatase ≤ 2.5 x ULN or ≤5x ULN if documented liver/bone metastases. Creatinine ≤ 1.5 ULN
    7. Blood urea within normal limits
11. Because of possible interference of cytochrome P450 3A4 activity by ixabepilone, patients were excluded from receiving the following medications at enrollment and while enrolled onto the study: amiodarone, clarithromycin, erythromycin, fluconazole, itraconazole, ketoconazole, indinavir, nelfinavir, ritonavir, and saquinavir
12. Women of childbearing age and potential must be willing to use effective contraception during the study and at least until 90 days after last dose of study drug. Male patients or male patients who have female partners of childbearing age and potential must be willing to use effective contraception during the study and at least until 90 days after last dose of study drug. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as intrauterine devices or hormonal contraception (oral contraceptive pills, implants, transdermal patches, vaginal rings or long-acting injections)

Exclusion Criteria:

1. HER2 positive tumor
2. Concurrent chemotherapy, radiotherapy, hormonal therapy, or other investigational drug except non-disease related conditions (e.g. insulin for diabetes) during study period
3. Patients with intracranial disease
4. Other malignancy with exception of curative treated non-melanoma skin cancer or cervical carcinoma in situ within 5 years prior to entering the study
5. Any active infection requiring parenteral or oral antibiotic treatment.
6. Patients with grade 2, in case of diabetes grade 1 or greater neuropathy
7. Clinically significant (i.e. active) cardiovascular disease:
8. Stroke within ≤ 6 months prior to day 1
9. Transient ischemic attach (TIA) within ≤ 6 months prior to day 1
10. Myocardial infarction within ≤ 6 months prior to day 1
11. Unstable angina
12. New York Hart Association (NYHA) Class II or greater congestive heart failure (CHF)
13. Serious cardiac arrhythmia requiring medication
14. Other medications or conditions, including surgery, that in the Investigator's opinion would contraindicate study participation for safety reasons or interfere with the interpretation of study results.
15. Requiring immediate palliative treatment of any kind including surgery and/or radiotherapy
16. Female patients who are pregnant or breast-feeding (pregnancy test with a positive result before study entry)
17. Known prior severe hypersensitivity reactions to agents containing polyoxyethylated castor oil (Cremophor EL)
18. Known hypersensitivity to fluoropyrimidines;
19. Known or suspected dihydropyrimidine dehydrogenase (DPD) deficiency;
20. Patients must not continue treatment with the following strong inhibitors of CYP3A4:

ketoconazole, itraconazole, ritonavir, amprenavir, indinavir, nelfinavir, delavirdine and voriconazole. These therapies should be discontinued 72 hours prior to initiation of study drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | 1 year
  To evaluate the clinical benefit rate of ixabepilone using tumor measurements (e.g. CT or MRI etc.). One-sided comparisons of CBR between treatment and historic control will be performed, and will be repeated for subgroups defined by ER status.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1 year
  PFS defined as time from inclusion until progressive disease(PD) according to RECIST v 1.0 or death of any reason
Overall survival (OS) | 1 year
  OS defined as time from inclusion until death
Overall response rate (ORR) defined as CR + PR | 1 year
  Objective response rate (ORR) as defined as complete response (CR) + partial response (PR) according to RECIST v 1.0
Incidence of Treatment-Emergent Adverse Events measured by NCI-CTCAE v.5.0 | 1 year
  A description of the extent, duration and reversibility of ixabepilone elicited toxicity in target organs based on the Common Terminology Criteria for Adverse Events (NCI-CTCAE v.5.0)
Clinical Benefit Rate (CBR) - fresh biopsy versus archival | 1 year
  Assess difference in prediction based on archival and fresh biopsy from same patient (percent agreement in binary prediction, and difference in primary and secondary endpoints with archival versus fresh biopsies)

CONTACTS AND LOCATIONS:
Locations (19):
- Belgium (4):
  - Antwerp University Hospital, Antwerp, Edegem
  - Onze-Lieve-Vrouwziekenhuis, Aalst
  - Clin. Univ. Saint-Luc, Brussels
  - CHU de Liege, Oncology Department, Liège
- Tampere University Hospital, Tampere, Finland
- Charité - Universitätsmedizin Berlin, Berlin, Germany
- Modena University Hospital, Modena, Italy
- Ikazia Hospital Rotterdam, Rotterdam, Netherlands
- Poland (4):
  - Wojewodzki Szpital Specjalietyczny, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii Ziemi Lubelskiej im., Lublin
  - Oddział Onkologii Klinicznej, Szpital Kliniczny Przemienienia Pańskiego UM w Poznaniu, Poznan
- United Kingdom (7):
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Somerset NHS Foundation Trust, Taunton, Somerset
  - Cancer Institute Singleton Hospital, Swansea, Wales
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh
  - St James Hospital, Leeds
  - Nottingham University Hospitals, Nottingham